CLINICAL TRIAL: NCT04553393
Title: Treatment of Decitabine-primed Tandem Targeting CD19 and CD20 Chimeric Antigen Receptor T Cells Plus Epigenetic Agents in Aggressive Relapsed and/or Refractory Non-Hodgkin's Lymphoma Patients With Huge Tumor Burden
Brief Title: Decitabine-primed Tandem CD19/CD20 CAR T Cells Plus Epigenetic Agents in Aggressive r/r B-NHL With Huge Tumor Burden
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-060
Record Dates: First submitted 2020-09-10; First posted 2020-09-17 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Refractory or Relapsed Aggressive r/r B-NHL With Huge Tumor Burden
MeSH Terms: interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; KPNA1 protein, human; Decitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Decitabine-primed Tandem CAR19/20 engineered T cells (Active Comparator): Tandem dual Specificity targeting CD19 and CD20 decitabine-primed CAR-T cells can recognize and kill the CD19 negative malignant cells through recognition of CD20 and improve the possibility of killing lymphoma tumor cells.
  Interventions: Biological: Decitabine-primed Tandem CAR19/20 engineered T cells
- Decitabine-primed Tandem CAR19/20 engineered T cells plus chidamide (Experimental): Chidamide is a novel and orally active benzamide class of HDAC inhibitor that selectively inhibits activity of HDAC1, 2, 3 and 10, which can Induce tumor-cell apoptosis, suppress cell proliferation and enhance immune surveillance.
  Interventions: Drug: Chidamide; Biological: Decitabine-primed Tandem CAR19/20 engineered T cells
- Decitabine-primed Tandem CAR19/20 engineered T cells plus decitabine (Experimental): Decitabine is an investigational (experimental) drug that works by depleting DNA methyltransferase 1(DNMT1), which can increase tumor antigens and HLA expression, enhances antigen processing, promotes T cell infiltration, and boosts effector T cell function.
  Interventions: Drug: Decitabine; Biological: Decitabine-primed Tandem CAR19/20 engineered T cells
- Decitabine-primed Tandem CAR19/20 engineered T cells plus chidamide+decitabine (Experimental): The combination of chidamide and decitabine can increase tumor antigens and HLA expression, enhances antigen processing, promotes T cell infiltration, and boosts effector T cell function, induce tumor-cell apoptosis, suppress cell proliferation and enhance immune surveillance
  Interventions: Drug: Chidamide and Decitabine; Biological: Decitabine-primed Tandem CAR19/20 engineered T cells

INTERVENTIONS:
Drug: Chidamide — Chidamide will be added 1 month after responding to CART cells infusion
  Other Names: cohort 2
  Arms: Decitabine-primed Tandem CAR19/20 engineered T cells plus chidamide
Drug: Decitabine — Decitabine will be added 1 month after responding to CART cells infusion
  Other Names: cohort 3
  Arms: Decitabine-primed Tandem CAR19/20 engineered T cells plus decitabine
Drug: Chidamide and Decitabine — Both chidamide and decitabine will be added 1 month after responding to CART cells infusion
  Other Names: cohort 4
  Arms: Decitabine-primed Tandem CAR19/20 engineered T cells plus chidamide+decitabine
Biological: Decitabine-primed Tandem CAR19/20 engineered T cells — Tandem CAR19/20 engineered T cells
  Other Names: cohort 1

SUMMARY:
This open-label, multi-cohorts, phase 1/2 study has the primary objective of comparing decitabine-primed tandem CART 19/20 solo, with decitabine-primed tandem CART 19/20 plus chidamide, decitabine-primed tandem CART 19/20 plus decitabine, and decitabine-primed tandem CART 19/20 plus decitabine+chidamide in patients with aggressive B-NHL who were confirmed as Relapsed and/or Refractory B cell Non-Hodgkin's Lymphoma with hugh tumor burden (Sum of the Product of the perpendicular Diameters for multiple lesions, SPD ≥ 100cm^2 or the largest-diameter of tumor ≥ 10 cm.).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥16 and ≤ 65 years.
2. Sum of the Product of the perpendicular Diameters for multiple lesions, SPD ≥ 100cm^2 or the largest-diameter of tumor ≥ 10cm.
3. Histologically confirmed CD20+ and/or CD19+ aggressive B-cell non-Hodgkin lymphoma (NHL), including the following types defined by the World Health Organization (WHO) 2016:

   * Diffuse large B-cell lymphoma (DLBCL).
   * High grade B-cell lymphoma(HGBL).
   * Other aggressive B-cell lymphoma.
4. Refractory disease or relapse after treatment with ≥2 lines of chemotherapy, including rituximab and anthracycline and either having failed autologous hematopoietic stem cell transplantation (HSCT), being ineligible for autologous HSCT or not consenting to autologous HSCT.

   We defined chemotherapy-refractory disease as meeting one or more of the following criteria:
   * No response to first-line therapy (primary refractory disease).
   * No response to second-line or later therapy.
   * Progressive disease (PD) as the best response to the most recent therapy regimen.
   * Stable disease (SD) as the best response after at least 2 cycles of the most recent line of therapy with an SD duration of no longer than 6 months from the last dose of therapy.

   Failure following autologous HSCT was defined as follows:
   * PD or relapsed disease ≤12 months after autologous stem cell transplantation (ASCT) (requires biopsy-proven recurrence in relapsed subjects).
   * No response or relapse after salvage therapy is given post-ASCT.
5. PD or relapse ≥3 months after treatment with targeted CD19 therapy, including CD19 CAR T cells or anti-CD19/anti-CD3.
6. Successful leukapheresis assessment and preculture of T cells.
7. Life expectancy > 3 months.
8. Adequate organ function:

   * Creatinine < 1.6 mg/dL (140 µmol/L) or creatinine clearance ≥60 mL/min.
   * Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) < 3× upper limit of the normal range.
   * Bilirubin <2.0 mg/dL unless the subject had Gilbert's syndrome (<3.0 mg/dL).
   * A minimum level of pulmonary reserve defined as ≤ grade 1 dyspnoea and pulse oxygenation > 91% with room air.
   * Cardiac ejection fraction ≥50%, no evidence of pericardial effusion as determined by an echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings.
9. An adequate bone marrow reserve defined as:

   * Absolute neutrophil count (ANC)>1,000/mm3.
   * Absolute lymphocyte count (ALC)≥300/mm3.
   * Platelet count ≥ 50,000/mm3.
   * Haemoglobin > 7.0 mg/dL.
10. Measurable or assessable disease according to the "IWG Response Criteria for Malignant Lymphoma" (Cheson 2014). Patients in complete remission (CR) with no evidence of disease were not eligible.
11. Informed consent/assent requiring that all patients have the ability to understand and the willingness to provide written informed consent.

Exclusion Criteria:

1. Patients with definite involvement of the gastrointestinal tract. Endoscopy should be performed to confirm gastrointestinal involvement in suspected patients. However, patients with central nervous system (CNS) involvement were cautiously enrolled in this clinical study.
2. Detection of a clear HAMA effect in patients with prior CD19 CAR T cell treatment failure or recurrence, or negative tumour puncture detection of CD19 and CD20.
3. Pregnant or lactating women.
4. Uncontrolled active bacterial or viral infection (active hepatitis B or hepatitis C infection, HIV infection) or treponema pallidum infection.
5. Class III/IV cardiovascular disability according to the New York Heart Association Classification and a cardiac ejection fraction ≥50%.
6. History of allo-HSCT.
7. Requirement for urgent therapy due to tumour mass effects such as respiratory obstruction or blood vessel compression.
8. Current or expected need for systemic corticosteroid therapy.
9. Any organ failure.
10. Patients with a second tumour requiring therapy or intervention.
11. Eastern Cooperative Oncology Group (ECOG) performance status score between 0 and 2.
12. Subjects considered unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation according to the investigator's judgement.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-09-08 (Estimated); Study Completion 2022-09-08 (Estimated)

PRIMARY OUTCOMES:
Adverse events after intervention | 12 months
  Safety Outcome
Progression Free Survival | 2 years
Duration of Response | 2 years
Overall Survival | 2 years

SECONDARY OUTCOMES:
Objective Response Rate Outcome Measure | 2 years
  ORR assess by investigators per the 2014 Lugano classification rate of subjects achieved objective response in all evaluable subjects
Intervention treatment-related adverse events (AEs) | 12 months
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0

OTHER OUTCOMES:
Exploratory research | 12 months
  Track cart cells in PB after infusions by TCR, transcriptional, and epigenetic sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, M.D., Principal Investigator — Chinese PLA Hospital
Locations (1):
- Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China